CLINICAL TRIAL: NCT04443530
Title: Evaluation of Effectiveness and Safety of Ultimaster™ Tansei™ Stent in Routine Clinical Practice; A Multicenter, Prospective Observational Study
Brief Title: Evaluation of Effectiveness and Safety of Ultimaster™ Tansei™ Stent in Routine Clinical Practice
Acronym: IRIS Tansei
Status: Recruiting | Type: Observational
Sponsor: Duk-Woo Park, MD (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Duk-Woo Park, MD, Associate Professor, Division of Cardiology, Asan Medical Center, University of Ulsan College of Medicine, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AMCCV2020-07
Record Dates: First submitted 2020-06-21; First posted 2020-06-23 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Coronary Artery Disease
Keywords: Tansei; Ultimaster; Ultimaster Tansei
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Coronary artery stenosis: Patients with coronary artery disease
  Interventions: Drug: Ultimaster™ Tansei™ stents

INTERVENTIONS:
Drug: Ultimaster™ Tansei™ stents — Patients receiving Ultimaster™ Tansei™ stents

SUMMARY:
This study is to evaluate the effectiveness and safety of Ultimaster Tansei stent in the "real-world" daily practice.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 19 years old
2. Patients receiving Ultimaster™ Tansei™ stents.
3. The patient or guardian agrees to the study protocol and the schedule of clinical follow-up and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethics Committee of the respective clinical site.

Exclusion Criteria:

1. Patients with a mixture of other drug-eluting stents (DESs)
2. Terminal illness with life-expectancy ≤1 year.
3. Patients with cardiogenic shock

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Ultimaster™ Tansei™ stents.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-09-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
The composite event rate of death, nonfatal myocardial infarction (MI), or ischemic-driven Target- Vessel Revascularization (TVR) | 1 year
  the composite of death, nonfatal myocardial infarction (MI), or ischemic-driven Target- Vessel Revascularization (TVR) at 12 months post-procedure.
  A composite endpoint is an endpoint that is a combination of multiple clinical endpoints. An event that is considered to have occurred if any one of several different events is observed.

SECONDARY OUTCOMES:
The event rate of all death | 5 years
The event rate of cardiac death | 5 years
The event rate of myocardial infarction | 5 years
The composite event rate of death or myocardial infarction | 5 years
the composite event rate of cardiac death or myocardial infarction | 5 years
The event rate of target-vessel revascularization | 5 years
The event rate of target-lesion revascularization | 5 years
The event rate of stent thrombosis | 5 years
  According to Academic Research Consortium(ARC) criteria
The event rate of stroke | 5 years
The event rate of procedural success | 3 days
  Defined as achievement of a final diameter stenosis of <30% by visual estimation, without the occurrence of death, Q-wave MI, or urgent revascularization during the index hospitalization.

CONTACTS AND LOCATIONS:
Locations (11):
- South Korea (11):
  - Gangwon National Univ. Hospital, Chuncheon
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - The Catholic University of Korea, Daejeon ST. Mary's Hospital, Daejeon
  - Gangneung Asan Hospital, Gangneung
  - Kwangju Christian Hospital, Kwangju
  - Pusan National University Hospital, Pusan
  - Asan Medical Center, Seoul
  - Kangdong Sacred Heart Hospital, Seoul
  - The Catholic Univ. of Korea Eunpyeong St. Mary's hospital, Seoul
  - St.Carollo Hospital, Suncheon

IPD SHARING:
Plan to Share IPD: Undecided